CLINICAL TRIAL: NCT05231044
Title: A Phase 3, Double-Blind, Vehicle-Controlled, Randomized, Parallel Group, Multicenter, Efficacy, Safety and PK Study of KX01 Ointment 1% in Japanese Adult Subjects With Actinic Keratosis on the Face or Scalp
Brief Title: A Multi-Center Study to Evaluate the Efficacy and Safety of KX01 Ointment 1% on Actinic Keratosis on Face or Scalp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Collaborators: PharmaEssentia Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B21-301
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Skin disease
MeSH Terms: conditions — Keratosis, Actinic; Skin Diseases

STUDY DESIGN:
Intervention Model Description: This study tests KX01 Ointment 1% against a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KX01 Ointment 1% (Experimental): KX01 Ointment 1% is applied topically once daily for 5 consecutive days on face or scalp
  Interventions: Drug: KX01 ointment 1%
- Placebo (Placebo Comparator): Vehicle Ointment is applied topically once daily for 5 consecutive days on face or scalp
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KX01 ointment 1% — The experimental drug, KX01 Ointment 1% is used in participants with Clinically typical AK on the face or scalp.
  Arms: KX01 Ointment 1%
Drug: Placebo — Vehicle Ointment is used in participants with Clinically typical AK on the face or scalp.
  Arms: Placebo

SUMMARY:
This Phase III study is designed to evaluate the efficacy and safety of KX01 Ointment in adult participants when applied to an area of skin containing more than 1, clinically typical Actinic Keratosis (AK) lesions on the face or scalp.

DETAILED DESCRIPTION:
This study is a double-blinded, multicenter, activity, and safety study of KX01 Ointment administered topically to the face or scalp of participants with actinic keratosis. The study consists of Screening, Treatment, Follow-up, and Recurrence Follow-up Periods. Eligible participants received 5 consecutive days of topical treatment, to be applied at the study site. Activity (lesion counts) and safety evaluations is performed.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese Males and females ≥20 years old
2. A treatment area on the face or scalp that:

   1. is a contiguous area measured 25 cm2
   2. contains more than 1 clinically typical, visible, and discrete AK lesions
3. Subjects who, in the judgment of the Investigator or Sub-investigator, are in good general health based on:

   1. medical history
   2. physical examination (PE) findings
   3. vital signs
   4. clinical chemistry, hematology, and urinalysis results
4. Females must be postmenopausal (>45 years of age with at least 12 months of amenorrhea), surgically sterile (by hysterectomy, bilateral oophorectomy, or tubal ligation); or, women with childbearing potential must use highly effective contraception for at least 30 days or 1 menstrual cycle, whichever is longer, prior to study treatment and must agree to continue to use highly effective contraception for at least 30 days following their last dose of study treatment. Highly effective contraception includes oral hormonal contraceptives, hormonal contraceptive implant, injection or patch, intrauterine device, or complete abstinence from sexual intercourse.
5. Sexually active males who have not had a vasectomy and whose partner is reproductively capable must agree to use barrier contraception from Screening until 90 days after their last dose of study treatment.
6. All subjects must agree not to donate sperm or eggs or attempt conception from Screening until 90 days following their last dose of study treatment.
7. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1 prior to randomization.
8. Willing to avoid excessive sunlight or ultraviolet (UV) light exposure, including the use of tanning beds, to the face or scalp

Exclusion Criteria:

1. Clinically atypical and / or rapidly changing AK lesions on the treatment area, e.g., hypertrophic, hyperkeratotic, recalcitrant disease (had cryosurgery on two previous occasions) and / or cutaneous horn
2. Location of the treatment area is:

   * On any location other than the face or scalp
   * Within 5 cm of an incompletely healed wound
   * Within 5 cm of a suspected basal cell carcinoma (BCC) or SCC
3. Been previously treated with KX01 Ointment
4. Anticipated need for in-patient hospitalization or in-patient surgery from Day 1 to Day 57
5. Treatment with 5-fluorouracil (5-FU), imiquimod, ingenol mebutate, diclofenac, photodynamic therapy, or other treatments for AK within the treatment area or within 2 cm of the treatment area, within 8 weeks prior to the Screening visit
6. Use of the following therapies and / or medications within 2 weeks prior to the Screening visit:

   * Cosmetic or therapeutic procedures (e.g., use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within the treatment area or within 2 cm of the selected treatment area
   * Acid-containing therapeutic products (e.g., salicylic acid or fruit acids, such as alpha- and beta-hydroxyl acids and glycolic acids), topical retinoids, or light chemical peels within the treatment area or within 2 cm of the selected treatment area
   * Topical salves (non-medicated / non-irritant lotion and cream are acceptable) or topical steroids within the treatment area or within 2 cm of the selected treatment area; artificial tanners within the treatment area or within 5 cm of the selected treatment area
7. Use of the following therapies and / or medications within 4 weeks prior to the Screening visit:

   * Treatment with immunomodulators (e.g., azathioprine), cytotoxic drugs (e.g., cyclophosphamide, vinblastine, chlorambucil, methotrexate), or interferons / interferon inducers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with complete (100%) clearance of Actinic Keratosis (AK) lesions | Day 57
  Complete clearance rate is defined as the percentage of participants at Day 57 with no clinically visible AK lesions in the treatment area.

SECONDARY OUTCOMES:
Partial Clearance Rate of AK Lesions at Day 57 | Day 57
  Partial clearance rate of AK lesions is defined as the proportion of subjects on Day 57 with a ≥ 75% reduction in the number of AK lesions identified at Baseline (Day 1 predose) in the treatment area.
Recurrence rate of AK lesions in subjects who achieved complete clearance at Day 57 | 3, 6, 9 and 12 months post-Day 57
  For subjects who achieve 100% clearance of AK lesions in the treatment area on Day 57, a Investigator or Sub-investigator will perform a count of clinically visible AK lesions (lesion count) during the Recurrence Follow-up Period at the 3-, 6-, 9- and 12-month visits. In principle, the Investigator or Sub-investigator performing the lesion count should be the same Investigator or Sub-investigator who evaluated the subject previously during the study.
Number of participants with local skin reactions (LSR) in the treatment area | Baseline (Day 1 predose), Days 5, 8, 15, 29 and 57
  At Baseline (Day 1 predose), LSRs on the treatment area will be assessed by the Investigator or Sub-investigator. The same Investigator or Sub-investigator will conduct the LSR assessment at all visits for an individual subject. LSR signs on the treatment area include the following: erythema, flaking / scaling, crusting, swelling, vesiculation / pustulation, and erosion / ulceration. These signs will be assessed using a 4-point grading scale.
Number of participants with pigmentation and scarring in the treatment area | Baseline (Day 1 predose), Days 5, 8, 15, 29 and 57
  At the time of LSR assessment, hypo- and hyper-pigmentation and scarring on the treatment area will be assessed by the Investigator or Sub-investigator as being present or absent. Pigmentation and scarring will be assessed at Baseline (Day 1 predose). In principle, the same Investigator or Sub-investigator will assess pigmentation and scarring at all visits for an individual subject.
Number of participants with Adverse Events (AEs), Serious Adverse Events (SAEs), events of special interest | From Baseline (Day 1 predose) up to Day 57
Number of participants with AEs within the treatment area after Day 57 up to 12 months post-Day 57 | After Day 57 up to 12 months post-Day 57

CONTACTS AND LOCATIONS:
Locations (20):
- Japan (20):
  - Toho University Medical Center Sakura Hospital, Chiba
  - Kiryu Dermatology Clinic, Fukuoka
  - Tomoko Matsuda dermatology Clinic, Fukuoka
  - Takamatsu Red Cross Hospital, Kagawa
  - Hashiguchi Dermatology, Kagoshima
  - Katahira Dermatology and Urology, Kagoshima
  - National Hospital Organization Sagamihara National Hospital, Kanagawa
  - Nippon Medical School Musashi Kosugi Hospital, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Noguchi Dermatology Clinic, Kumamoto
  - Suizenji Dermatology Clinic, Kumamoto
  - Futaba Dermatology and Skin Surgery Clinic, Miyazaki
  - Toyama Hifuka, Miyazaki
  - Okayama Saiseikai Outpatient Center Hospital, Okayama
  - Medical Corporation Ayumi Sakurakai Dermatology Ophthalmology Kume Clinic, Osaka
  - Mochidahifuka, Osaka
  - Juntendo University Hospital, Tokyo
  - NTT Medical Center Tokyo, Tokyo
  - Toyama Prefectural Central Hospital, Toyama
  - University of Yamanashi Hospital, Yamanashi